CLINICAL TRIAL: NCT01378689
Title: Improving Bone Health Among RA Patients on Chronic Glucocorticoids
Brief Title: Improving Bone Health Among Rheumatoid Arthritis (RA) Patients on Chronic Glucocorticoids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Medco Health Services, Inc (Unknown)
Responsible Party: Principal Investigator, Kenneth Saag, MD, MSc, Jane Knight Lowe Professor of Medicine, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: X080529001
Record Dates: First submitted 2011-06-16; First posted 2011-06-22 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Adverse Effect of Glucocorticoids and Synthetic Analogues; Osteoporosis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoporosis; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online video (Experimental): Participants in this arm are shown a brief video (~5 minutes) after ordering a refill for their glucocorticoid use. The video includes real patients telling their own story about the possible side effects of prolonged use of glucocorticoids.
  Interventions: Other: Storytelling online video
- No video (No Intervention)

INTERVENTIONS:
Other: Storytelling online video — patients with a history of chronic glucocorticoids use tell their experiences of side effects resulting from chronic use and provide advice on ways to prevent side effects
  Arms: Online video

SUMMARY:
This quality improvement project is aimed at improving health care by identifying low cost strategies to get Rheumatoid Arthritis (RA) patients to more effectively communicate with their physicians about osteoporosis prevention and treatment (improving doctor-patient communication). The investigators will implement a direct to patient intervention to the population of interest (patients on chronic glucocorticoids) via story-telling, using an Internet based video. The target audience is people on chronic glucocorticoids not already receiving bones-specific osteoporosis medications to determine differences in post-intervention rates of osteoporosis care, and the rates of prescription anti-osteoporosis therapies.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 5 milligrams of prednisone or glucocorticoid dose equivalent for greater than or equal to 90 days within the previous 12 months
* Medco member for entire study period
* Refill steroid prescription online

Exclusion Criteria:

* anti-osteoporosis medication in previous 12 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4659 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of participants receiving Anti-osteoporosis Treatment | within 3 - 12 months of exposure to video
  Includes bisphosphonates, PTH, SERM, Calcitonin

SECONDARY OUTCOMES:
Calcium and Vitamin D use | within 3 - 12 months of exposure to video
  Are participants taking calcium and vitamin d supplements
Patient-Physician Communication | within 3 - 12 months of exposure to video
  Did viewing the video increase patient-physician communication

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Saag, MD, MSc, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Warriner AH, Outman RC, Allison JJ, Curtis JR, Markward NJ, Redden DT, Safford MM, Stanek EJ, Steinkellner AR, Saag KG. An Internet-based Controlled Trial Aimed to Improve Osteoporosis Prevention among Chronic Glucocorticoid Users. J Rheumatol. 2015 Aug;42(8):1478-83. doi: 10.3899/jrheum.141238. Epub 2015 Jul 1. PMID 26136484